CLINICAL TRIAL: NCT03929666
Title: Phase 2 Study of ZW25 Plus First-line Combination Chemotherapy in HER2-Expressing Gastrointestinal (GI) Cancers, Including Gastroesophageal Adenocarcinoma (GEA), Biliary Tract Cancer (BTC), and Colorectal Cancer (CRC)
Brief Title: A Safety and Efficacy Study of ZW25 (Zanidatamab) Plus Combination Chemotherapy in HER2-expressing Gastrointestinal Cancers, Including Gastroesophageal Adenocarcinoma, Biliary Tract Cancer, and Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW25-201
Expanded Access: NCT04578444 (No longer available)
Record Dates: First submitted 2019-02-22; First posted 2019-04-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: HER2-expressing Gastrointestinal Cancers, Including Gastroesophageal Adenocarcinoma, Biliary Tract Cancer, and Colorectal Cancer
Keywords: HER2; Bispecific antibody; Biparatopic antibody; Immunotherapy; Gastric cancers; Esophageal cancers; Gastroesophageal junction (GEJ) cancers; Chemotherapy; FP; mFOLFOX6; Capecitabine; Cisplatin; 5-FU; Leucovorin (folinic acid); Oxaliplatin; XELOX; Gastrointestinal cancers; Gastroesophageal adenocarcinoma; Biliary tract cancer; Colorectal cancer; Intrahepatic cholangiocarcinoma; Extrahepatic cholangiocarcinoma; Gall bladder
MeSH Terms: conditions — Biliary Tract Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Neoplasms; Gastrointestinal Neoplasms; Cholangiocarcinoma | interventions — zanidatamab; Capecitabine; Cisplatin; Fluorouracil; Leucovorin; Oxaliplatin; Bevacizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ZW25 + FP (Experimental): ZW25 plus fluorouracil (5-FU) and cisplatin
  Interventions: Drug: ZW25 (Zanidatamab); Drug: Cisplatin; Drug: Fluorouracil
- ZW25 + mFOLFOX6 (Experimental): ZW25 plus 5-FU, leucovorin, and oxaliplatin
  Interventions: Drug: ZW25 (Zanidatamab); Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- ZW25 + XELOX (Experimental): ZW25 plus capecitabine and oxaliplatin
  Interventions: Drug: ZW25 (Zanidatamab); Drug: Capecitabine; Drug: Oxaliplatin
- ZW25 + mFOLFOX6 with bevacizumab (Experimental): ZW25 plus 5-FU, leucovorin, oxaliplatin, and bevacizumab
  Interventions: Drug: ZW25 (Zanidatamab); Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Bevacizumab
- ZW25 + CisGem (Experimental): ZW25 plus cisplatin and gemcitabine
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: ZW25 (Zanidatamab) — * Part 1: administered IV at dose levels and schedules determined by the Safety Monitoring Committee (SMC)
  * Part 2: RD identified in Part 1
  Arms: ZW25 + FP; ZW25 + XELOX; ZW25 + mFOLFOX6; ZW25 + mFOLFOX6 with bevacizumab
Drug: Capecitabine — Administered orally twice daily (PO bid)
  Arms: ZW25 + XELOX
Drug: Cisplatin — Administered IV
  Arms: ZW25 + CisGem; ZW25 + FP
Drug: Fluorouracil — Administered IV
  Arms: ZW25 + FP; ZW25 + mFOLFOX6; ZW25 + mFOLFOX6 with bevacizumab
Drug: Leucovorin — Administered IV
  Arms: ZW25 + mFOLFOX6; ZW25 + mFOLFOX6 with bevacizumab
Drug: Oxaliplatin — Administered IV
  Arms: ZW25 + XELOX; ZW25 + mFOLFOX6; ZW25 + mFOLFOX6 with bevacizumab
Drug: Bevacizumab — Administered IV
  Arms: ZW25 + mFOLFOX6 with bevacizumab
Drug: Gemcitabine — Administered IV
  Arms: ZW25 + CisGem

SUMMARY:
This is a multicenter, global, Phase 2, open-label, 2-part, first-line study to investigate the safety, tolerability, and anti-tumor activity of ZW25 (zanidatamab) plus standard first-line combination chemotherapy regimens for selected gastrointestinal (GI) cancers. Eligible patients include those with unresectable, locally advanced, recurrent or metastatic HER2-expressing gastroesophageal adenocarcinoma (GEA), biliary tract cancer (BTC), or colorectal cancer (CRC).

DETAILED DESCRIPTION:
Part 1 of the study will first evaluate the safety and tolerability of ZW25 plus standard first-line combination chemotherapy (XELOX, FP, or mFOLFOX6 for GEA; mFOLFOX6 with or without bevacizumab for CRC; and CisGem for BTC) and will confirm the recommended dosage (RD) of ZW25 when administered in combination with each of these multi-agent chemotherapy regimens. Then, Part 2 of the study will evaluate the anti-tumor activity of ZW25 plus combination chemotherapy in HER2-expressing GEA, BTC, and CRC.

ELIGIBILITY:
Inclusion:

* Disease diagnosis:

  * Part 1:
  * GEA: Unresectable, locally advanced, recurrent or metastatic HER2-expressing GEA (IHC 3+ or 2+ with or without gene amplification based upon local assessment or central assessment)
  * BTC: Unresectable, locally advanced, recurrent or metastatic HER2-expressing BTC (including intrahepatic cholangiocarcinoma [ICC], extrahepatic cholangiocarcinoma [ECC], or gallbladder cancer [GBC]) (IHC 3+ with or without gene amplification; or IHC 0, 1+ or 2+ with gene amplification, based upon central assessment)
  * CRC: Unresectable, locally advanced, recurrent or metastatic HER2-expressing CRC (IHC 3+ with or without gene amplification; or IHC 0, 1+ or 2+ with gene amplification, based upon central assessment). Patients will be required to be extended RAS (KRAS and NRAS) and BRAF wild-type based upon central assessment.
  * Part 2:
  * GEA: Unresectable, locally advanced, recurrent or metastatic HER2-expressing GEA (IHC 3+, or IHC 2+ and FISH+ by central assessment)
  * BTC: Same as Part 1
  * CRC: Same as Part 1
* Tumor measurements as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1:

  * Part 1: Measurable or non-measurable disease
  * Part 2: Measurable disease
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Adequate organ function
* Adequate cardiac left ventricular function, as defined by a LVEF >/= institutional standard of normal

Exclusion:

* Prior treatment with a HER2-targeted agent
* Prior systemic anti-cancer therapy (including investigational products) except prior adjuvant/neoadjuvant therapy, which must be completed at least 6 months prior to first study treatment dosing. For subjects with BTC and CRC the following additional exceptions apply:

  * BTC: patients may have started therapy for advanced disease but may not have received more than one cycle of any standard gemcitabine-based chemotherapy regimen.
  * CRC: patients may have started therapy for advanced disease but may not have received more than one cycle of 5-FU-based chemotherapy (< 1 month of therapy).
* Patients with certain contraindications to bevacizumab cannot be enrolled on the mFOLFOX6-2 with bevacizumab arm.
* Palliative radiotherapy is allowed if completed at least 2 weeks prior to first study treatment dosing
* Untreated known brain metastases (patients with treated brain metastases who are off steroids, off antiseizure medications, and stable for at least 1 month at the time of screening are eligible)
* Clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension or any history of symptomatic congestive heart failure (CHF). Patients with known myocardial infarction or unstable angina within 6 months prior to randomization are also excluded.
* QTc Fridericia (QTcF) > 470 ms. For patients with longer QTcF on initial electrocardiogram (ECG), follow-up ECG may be performed in triplicate to determine eligibility
* Peripheral neuropathy > Grade 1 per NCI-CTCAE v5.0
* Clinically significant interstitial lung disease
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Active hepatitis B or hepatitis C infection or infection with Human Immunodeficiency Virus (HIV)-1 or HIV-2 (Exception: patients with well controlled HIV [e.g., CD4 > 350/mm3 and undetectable viral load] are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) (Part 1) | Up to 6 weeks
  Number of participants who experienced a DLT. DLTs include adverse events considered to be related to study treatment, including the evaluated dose level of ZW25, any component or combination of the components of a chemotherapy regimen, or the combination of ZW25 plus a chemotherapy regimen.
Incidence of adverse events (Part 1) | Up to 11 months
  Number of participants who experienced an adverse event
Incidence of lab abnormalities (Part 1) | Up to 11 months
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology and chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Objective response rate (ORR) (Part 2) | Up to 10 months
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) (Part 1) | Up to 10 months
  Number of participants who achieved a best response of either CR or PR during treatment per RECIST 1.1
Disease control rate (Parts 1 and 2) | Up to 10 months
  Number of participants who achieved a best response of CR, PR, or stable disease (SD) during treatment per RECIST 1.1
Duration of response (Parts 1 and 2) | Up to 2 years
  Median duration of response (in months) and range (minimum, maximum)
Clinical benefit rate (Parts 1 and 2) | Up to 2 years
  Number of participants with SD for ≥ 24 weeks or a confirmed, best overall response of CR or PR per RECIST 1.1
Progression-free survival (Parts 1 and 2) | Up to 2 years
  Median progression-free survival (in months) and range (minimum, maximum)
Overall survival (Parts 1 and 2) | Up to 2 years
  Median overall survival (in months) and range (minimum, maximum)
Incidence of anti-drug antibodies (ADAs) (Parts 1 and 2) | Up to 11 months
  Number of participants who develop ADAs
End of infusion concentration of ZW25 (Parts 1 and 2) | Up to 11 months
Maximum serum concentration of ZW25 (Parts 1 and 2) | Up to 11 months
Trough concentration of ZW25 (Parts 1 and 2) | Up to 11 months
Incidence of adverse events (Part 2) | Up to 11 months
  Number of participants who experienced an adverse event
Incidence of lab abnormalities (Part 2) | Up to 11 months
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology and chemistry. Grades are defined using National Cancer Institute's CTCAE, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Garfin, MD, PhD, Study Director — Jazz Pharmaceuticals
Locations (23):
- United States (11):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - The Cancer and Hematology Centers, Grand Rapids, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Chile (4):
  - Centro de Investigacion Clinica SAGA, Santiago
  - Icegclinic Research & Care, Santiago
  - CECIM Biocinetic, Santiago
  - Centro Internacional de Estudios Clínicos, Santiago
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University, Busan
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elimova E, Ajani J, Burris H, Denlinger CS, Iqbal S, Kang YK, Kim JH, Lee KW, Lin B, Mehta R, Oh DY, Rha SY, Seol YM, Yang L, Ozog MA, Garfin PM, Ku G. Zanidatamab plus chemotherapy as first-line treatment for patients with HER2-positive advanced gastro-oesophageal adenocarcinoma: primary results of a multicentre, single-arm, phase 2 study. Lancet Oncol. 2025 Jul;26(7):847-859. doi: 10.1016/S1470-2045(25)00287-6. Epub 2025 Jun 2. PMID 40473445